CLINICAL TRIAL: NCT04642859
Title: Training Second-grade Dyslexic Students Using a Computerized Program in Assiut, Egypt
Acronym: Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Osama Aboshaera, Associate Professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU Dyslexia
Record Dates: First submitted 2020-11-12; First posted 2020-11-24 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Dyslexia
Keywords: Dyslexia; Training; Egypt
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: compare scores before and after the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dyslexia (Experimental): Students with dyslexia before and after the intervention
  Interventions: Behavioral: Computerized Cognitive abilities training battery for reading (CATB-R)

INTERVENTIONS:
Behavioral: Computerized Cognitive abilities training battery for reading (CATB-R) — Specially designed Arabic computerized training program for dyslexia

SUMMARY:
Dyslexia is a specific learning disability that is neurological in origin. It is characterized by difficulties with accurate or fluent word recognition, by poor spelling and decoding abilities, difficulty reading words in isolation and difficulty with oral reading (slow, inaccurate, or labored). These difficulties typically result from a deficit in the phonological component of language that is often unexpected with other cognitive abilities and the provision of effective classroom instruction. The phonological deficit hypothesis is the dominant explanatory theory of developmental dyslexia. Despite this, impaired phonological processing alone cannot explain all clinical symptoms of dyslexia. Many students with dyslexia have multiple deficits other than phonological deficits. Of these accused deficits are visual perceptual processing deficits, auditory processing deficits, multisensory spatial attention deficits as well as cerebellar dysfunction. The current mandatory criterion for the diagnosis of dyslexia, below-average achievement, implies waiting to failure. This approach for diagnosis (must fail approach) would delay intervention for rehabilitation.

Furthermore, the cut-off scores would result in over or under inclusion of cases and appear to be the least reliable and valid approach to diagnosis. Both methods lack a deeper understanding of the underlying reading difficulty, their neurobiological basis, and hence represent barriers against scientifically-based interventions. However, improved understanding of the neurobiological basis of dyslexia will facilitate evidence-based effective intervention.

DETAILED DESCRIPTION:
This study will be carried out along seven stages; 1- Identification of students with reading disability using Arabic Reading Achievement test (RAT); 2- Construction of a computerized Arabic Cognitive Abilities diagnostic battery for Reading (CADB-R); 3- Standardization of the constructed battery; 4- Detailed study of the cognitive profile; 5- Construction of a Computerized Cognitive abilities training battery for reading (CATB-R); 6- Application of the training battery; 7- Reassessment.

ELIGIBILITY:
Inclusion Criteria:

* 2nd-grade primary school students
* Poor scholastic achievement: less than mean - SD score on Arabic reading achievement test
* Normal neurological, basic audiological, and ophthalmological examination
* Both sexes included

Exclusion Criteria:

* Student refused to participate
* Abnormal neurological, audiological or ophthalmological examination

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Arabic Reading Achievement test (RAT) | Baseline, 2 months
  new scale of Arabic Reading Achievement test specially designed for this study. Students will classified according to their achievement level into three groups:
  1. Group I: Poor achievers (scores < mean - SD), considered students with reading disability, or dyslexia
  2. Group II: Average achievers (with scores= mean + SD)
  3. Group III included those with good achievement (score > mean+ SD)

SECONDARY OUTCOMES:
Change in Computerized Arabic Cognitive Abilities diagnostic battery for Reading (CADB-R) | Baseline, 2 months
  Specially designed battery in a game-like manner to test a wide range of cognitive skills that are supposed to be important in the early stages of learning to read. It includes the following skills:
  1. Text Reading comprehension
  2. Visual discrimination
  3. Auditory discrimination
  4. Phonological awareness
  5. Visuospatial skills
  6. Audio-Visual correspondence
  7. Auditory memory

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M Farghaly, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt